CLINICAL TRIAL: NCT03802604
Title: Combination of Talimogene Laherparepvec With Atezolizumab in Patients With Residual Breast Cancer After Standard Neoadjuvant Multi-agent Chemotherapy (PROMETEO TRIAL)
Brief Title: Combination of Talimogene Laherparepvec With Atezolizumab in Early Breast Cancer
Acronym: PROMETEO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Amgen (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1503; 2018-001300-10 (EudraCT Number)
Record Dates: First submitted 2018-11-15; First posted 2019-01-14 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: atezolizumab; T-vec; talimogene laherparepvec
MeSH Terms: conditions — Breast Neoplasms | interventions — talimogene laherparepvec; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Talimogene laherparepvec + Atezolizumab (Experimental): 1. Talimogene laherparepvec: Cycle 1 - 10^6 PFU/mL. Cycle 2, 3, 4 & 5 - 10^8 PFU/mL.
  2. Atezolizumab 840 mg
  Interventions: Biological: Talimogene laherparepvec; Drug: Atezolizumab

INTERVENTIONS:
Biological: Talimogene laherparepvec — Talimogene laherparepvec will be given via intra-tumoral injection at an initial dose of 10^6 PFU/mL. On week 3 (i.e. 21 days [± 2] days), a second talimogene laherparepvec injection will be administered at a dose of 10^8 PFU/mL. Third, fourth and fifth injections will be administered every 2 weeks (every 14 [± 2] days). The maximum volume for each injection will be 4.0 mL.
  Other Names: T-VEC; Imlygic
Drug: Atezolizumab — Atezolizumab 840 mg will be administered by IV infusion on Day1 week 3, then every 2 weeks (every 14 [± 2] days), for a total of 4 treatment courses.
  Other Names: Tecentric

SUMMARY:
PROMETEO is a window opportunity, single arm, exploratory study to evaluate the effect of T- VEC combined with Atezolizumab in women with operable early breast cancer who present residual disease after Neoadjuvant Chemotherapy (NAC). Other eligibility criteria include TNBC or LumB like primary tumor sized at least 1.5 cm, ECOG PS 0-1 and evaluable diagnostic tumor sample.

DETAILED DESCRIPTION:
Primary objective:

• To evaluate the efficacy (as measured by residual cancer burden [RCB] class 0/1 rate) of Talimogene Laherparepvec with Atezolizumab given to subjects with operable early breast cancer who present residual disease after neoadjuvant chemotherapy (NAC).

Secondary objectives include:

* To assess the rate of pathological complete response (pCR) in the breast (pCRB) and breast and axilla (pCRBL) at definitive surgery after neoadjuvant treatment with T-VEC and atezolizumab.
* To determine the clinical and radiological ORR of breast tumors to TVEC- atezolizumab given in the neoadjuvant setting.
* To assess RCB index in continuous variable and by the 4 RCB class (RCB0, RCB1, RCB2 and RCB 3) after treatment with T-VEC and atezolizumab.
* Comparing the expression of a gene signature tracking activated CD8 T-cells at surgery after treatment with T-VEC and atezolizumab with residual disease after NAC.
* To evaluate the safety of T-VEC in combination with atezolizumab as assessed by incidence of treatment-emergent and treatment-related adverse events.
* Translational and exploratory objectives are included.

ELIGIBILITY:
Patient inclusion criteria

1. Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
2. Female patients age ≥18 years at the time of informed consent.
3. Histologically confirmed diagnosis of non-metastatic primary invasive adenocarcinoma of the breast, with all of the following characteristics:

   * TNBC or luminal B-like/HER2-negative breast cancer.
   * At least 1 lesion that can be accurately and serially measured in at least 1 dimension and for which the longest diameter is ≥ 10 mm as measured by magnetic resonance imaging (MRI).
   * Breast cancer eligible for primary surgery
   * In the case of a multifocal/multicentric tumor, the largest lesion must be ≥ 15 mm and designated the "target" lesion for all subsequent tumor evaluations.
4. ER, PgR and HER2 tumor determination by ASCO/CAP guidelines locally assessed:

   * TNBC defined as: ER and PR negative defined as IHC nuclear staining <1% AND HER2 negative.
   * Luminal B-like/HER2 negative defined as:

     * ER or PR positive defined as IHC nuclear staining ≥1% AND HER2 negative AND local Ki-67 ≥20% or
5. Patient must have injectable and biopsiable disease (direct injection or ultrasound guided).
6. Completed ≥ 80% total dose of an anthracycline/taxane-based neoadjuvant regimen recommended by the NCCN guidelines. The addition of carboplatin to a taxane is allowed.
7. ECOG Performance Status of 0 or 1.
8. Adequate organ function determined within 14 days prior to enrollment, defined as follows:

   * Hematological

     * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
     * Platelet count ≥ 100 x 109/L
     * Hemoglobin ≥ 9 g/dL (red blood cell transfusion and/or erythropoietin allowed)
   * Renal

     o Serum creatinine ≤ 1.5 x upper limit of normal (ULN), or 24-hour creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN. (Note: Creatinine clearance does not need to be determined if the baseline serum creatinine is within normal limits. Creatinine clearance should be calculated per institutional standard).
   * Hepatic

     * serum bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN
     * aspartate aminotransferase (AST) ≤ 2.5 x ULN alanine aminotransferase (ALT) ≤ 2.5 x ULN
     * Coagulation International normalization ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN
9. Partial thromboplastin time (PTT) or activated PTT (aPTT) ≤ 1.5 x ULN
10. Absence of any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule; those situations should be discussed with the patient before registration in the trial.
11. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 4.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion).

Patient exclusion criteria

1. Inoperable locally advanced breast cancer after NAC.
2. Metastatic (Stage IV) breast cancer.
3. Bilateral invasive breast cancer.
4. Prior therapy with an anti- PD-1, anti- PD-L1, anti-PD-L2, anti-CD137 antibody, or anti-CTLA- 4 antibody compound, T-VEC or any other oncolytic immunotherapy.
5. Prior therapy with tumor vaccine.
6. Currently receiving treatment in another investigational device or study drug, or less than 28 days since ending treatment on another investigational device or study drug.
7. History or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease, or active autoimmune disease or syndrome that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). with the following exceptions:

   * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
   * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

   Rash must cover 10% of body surface. Disease is well controlled at baseline and requires only low-potency topical corticosteroids.

   No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
8. Active herpetic skin lesions or prior complications of herpetic infection (e.g. herpetic keratitis or encephalitis) and must not require intermittent or chronic treatment with an antiherpetic drug (e.g. acyclovir), other than intermittent topical use.
9. Received live vaccine within 28 days prior to enrollment or within 5 months after the last dose of atezolizumab.
10. Evidence of clinically significant immunosuppression such as the following:

    * diagnosis of immunodeficiency
    * concurrent opportunistic infection
    * receiving systemic immunosuppressive therapy (> 2 weeks) or within 7 days prior to the first dose of study treatment, including oral steroid doses > 10 mg/day of prednisone or equivalent. Subjects that require intermittent use of bronchodilators or local steroid injection will not be excluded from the study.
11. Cardiopulmonary dysfunction as defined by:

    * Uncontrolled hypertension (systolic >150 mm Hg and/or diastolic > 100 mm Hg) despite optimal medical management.
    * Inadequately controlled angina or serious cardiac arrhythmia not controlled by adequate medication.
    * History of symptomatic congestive heart failure (CHF): Grade ≥ 3 per NCI CTCAE version 4.0 or Class ≥ II New York Health Association (NYHA criteria).
    * Myocardial infarction within 6 months prior to enrollment.
    * Current dyspnea at rest due to complications of advanced malignancy, or other disease requiring continuous oxygen therapy
12. Current severe, uncontrolled systemic disease (e.g. clinically significant cardiovascular, pulmonary or metabolic disease; wound healing disorders; ulcers; bone fractures).
13. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
14. Uncontrolled or symptomatic hypercalcemia (ionized calcium 1.5 mmol/L, calcium 12 mg/dL or corrected serum calcium ULN)
15. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
16. Major surgical procedure or significant traumatic injury within approximately 28 days prior to enrollment or anticipation of the need for major surgery during the course of study treatment.
17. Concurrent, serious, uncontrolled infections or current known infection with HIV or active hepatitis B and/or hepatitis C.
18. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment with exception of prophylactic antibiotics
19. Has a known history of active Bacillus tuberculosis
20. Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of talimogene laherparepvec or 5 months after the last dose of atezolizumab, whichever is later
21. Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec or 5 months after the last dose of atezolizumab, whichever is later. Note: Women not of childbearing potential are defined as:

    * postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.) OR
    * have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening; OR
    * has a congenital or acquired condition that prevents childbearing.

    Note: Acceptable methods of effective contraception are defined in the informed consent form and Appendix A.
22. Subject has known sensitivity to any of the products or components to be administered during dosing
23. Assessment by the investigator to be unable or unwilling to comply with the requirements of the protocol.
24. History of other malignancy within 5 years prior to screening, except for appropriately treated basal or squamous cell carcinoma, carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer.
25. History of significant co-morbidities that, in the judgment of the investigator, may interfere with the conduction of the study, the evaluation of response, or with informed consent.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Rate of residual cancer burden class 0 and 1 (RCB0/1) | 24 months since first patient in
  As a dichotomous measure of tumor response, RCB 0/1 yes vs. no., after neoadjuvant treatment, according to the MD Anderson Cancer Center procedures, as per local assessment.

SECONDARY OUTCOMES:
Rate of pCRB (ypT0/Tis) and pCRBL (ypT0/TisypN0) | 24 months since first patient in
  Complete absence of invasive carcinoma in the breast or in the breast and axillary lymph nodes on histological examination at the time of definitive surgery, irrespective of in situ carcinoma in the breast and in the breast and axilla by local evaluation will be assessed.
Tumor ORR | 24 months since first patient in
  Defined as the sum of PR and CR according to RECIST v1.1, as per Investigator's assessments by breast MRI.
Rate of residual cancer burden (RCB) | 24 months since first patient in
  As a continuous variable and by RCB group, after neoadjuvant treatment, according to the MD Anderson Cancer Center procedures, as per local assessment.
Changes in the expression of a gene signature tracking activated CD8 T-cells. | 24 months since first patient in
  Differences in in the mean expression of an immune gene signature tracking CD8 T-cells (composed of the following genes: PRF1, CD8A, GZMM, CD8B, FLT3LG) in all patients will be assessed.
Incidence, duration and severity of AEs assessed by the NCI Common Terminology for Classification of Adverse Events (CTCAE) version 4 | 24 months since first patient in
  Incidence, duration and severity of AEs assessed by the NCI Common Terminology for Classification of Adverse Events (CTCAE) version 4, including delays and treatment discontinuations.

CONTACTS AND LOCATIONS:
Overall Officials: Aleix Prat, Principal Investigator — Hospital Clinic of Barcelona
Locations (4):
- Spain (4):
  - Hospital Universitari Vall d'Hebrón, Barcelona, Barcelona
  - Centro Integral Oncológico Clara Campal, Madrid, Madrid
  - Hospital Clínico universitario de Valencia, Valencia, Valencia
  - Hospital Clínic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pascual T, Cejalvo JM, Oliveira M, Vidal M, Vega E, Ganau S, Julve A, Zamora E, Miranda I, Delgado A, Bermejo B, la Cruz-Merino L, Juan M, Ferrero-Cafiero JM, Canes J, Gonzalez X, Villagrasa P, Prat A. SOLTI-1503 PROMETEO TRIAL: combination of talimogene laherparepvec with atezolizumab in early breast cancer. Future Oncol. 2020 Aug;16(24):1801-1813. doi: 10.2217/fon-2020-0246. Epub 2020 Jul 7. PMID 32633563